CLINICAL TRIAL: NCT00991796
Title: Randomised, Double-Blinded, Placebo Controlled, Phase 2 Study of CS-1008 in Combination With Carboplatin/Paclitaxel in Chemotherapy naïve Subjects With Metastatic or Unresectable Non-small Cell Lung Cancer
Brief Title: CS-1008 With Carboplatin/Paclitaxel in Chemotherapy naïve Subjects With Metastatic or Unresectable Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS1008-A-E202
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tigatuzumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS-1008 (Experimental): CS-1008 with carboplatin and paclitaxel
  Interventions: Drug: CS-1008; Drug: Paclitaxel; Drug: Carboplatin
- Placebo (Placebo Comparator): Placebo with carboplatin and paclitaxel
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: CS-1008 — CS-1008 powder for concentrate for solution for infusion. six cycles of combination therapy with 3 weeks equal to one cycle. 10 mg/kg
  Arms: CS-1008
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Paclitaxel — Paclitaxel concentrate for solution for infusion. once every 3 weeks for a maximum of 6 cycles. 175 mg/m2
  Other Names: Taxol
Drug: Carboplatin — Carboplatin concentrate for solution for infusion. once every 3 weeks for a maximum of 6 cycles. 6 mg/m2
  Other Names: Paraplatin

SUMMARY:
The purpose of this study is to determine the effect on toxicity of the addition of CS 1008 to a platinum based chemotherapy regimen on the progression-free survival (PFS) in subjects with stage IIIB wet or stage IV NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Measurable disease as defined by RECIST criteria
* Adequate organ and bone marrow function as evidenced by:

  * Hemoglobin >= 9 g/dL;
  * ANC >= 1.5 x 109/L;
  * Platelet count >= 100 x 109/L;
  * Serum creatinine < 1.5 mg/dL or creatinine clearance > 60 mL/min;
  * AST, ALT, and alkaline phosphatase <= 2.5 x upper limit of normal (ULN) if without liver metastasis and <= 5.0 x ULN if liver metastasis;
  * Total bilirubin <= 2.0 x ULN.
* Men and women of childbearing potential must be willing to consent to using effective double barrier contraception (eg, hormonal contraceptives, bilateral tubal ligation, barrier with spermicidal, intrauterine device) while on treatment and for 3 months thereafter.
* All female subjects of childbearing potential must have a negative pregnancy test (serum or urine) result <= 72 hours before initiating study treatment.
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IEC approved ICF before performance of any study specific procedures or tests.

Exclusion Criteria:

* Anticipation of need for a major surgical procedure or radiotherapy (RT) during the study.
* Prior treatment with chemotherapy for their disease.
* History of any of the following conditions within 6 months before study enrolment: myocardial infarction; New York Heart Association (NYHA) class II or higher severe/unstable angina pectoris; coronary/peripheral artery bypass graft; NYHA class III or IV congestive heart failure; cerebrovascular accident or transient ischemic attack, pulmonary embolism, or other clinically significant thromboembolic event; clinically significant pulmonary disease (eg, severe chronic obstructive pulmonary disease or asthma); clinically significant pulmonary edema or anasarca.. See Section 17.2 for NYHA Classification.
* Clinically significant pleural or pericardial effusions.
* Grade 2 or higher current peripheral neuropathy (See Section 17.3; NCI CTCAE, Version 3.0).
* Clinically active brain metastasis (ie, untreated, still requiring therapy with steroids or RT, or with progression within 4 weeks after completion of RT); an uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis.
* History of malignancy other than NSCLC, unless there is the expectation that the malignancy has been cured, and tumor specific treatment for the malignancy has not been administered within the previous 5 years.
* Clinically significant active infection that requires antibiotic therapy or Human Immunodeficiency Virus (HIV) positive subjects receiving antiretroviral therapy.
* Previous treatment with chemotherapy, CS 1008, other agonistic DR 5 or DR 4 antibodies, or with TRAIL.
* Pregnant or breast feeding.
* Known history of hypersensitivity reactions to any of the components of CS 1008, carboplatin, or paclitaxel formulations.
* Serious intercurrent medical or psychiatric illnesses or any other conditions that in the opinion of the Investigator would impair the ability to give informed consent or unacceptably reduce protocol compliance or safety of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Difference in progression-free survival (PFS) of patients treated with CS-1008 and paclitaxel/carboplatin versus placebo and paclitaxel/carboplatin | 6 months

SECONDARY OUTCOMES:
Difference in overall survival of patients treated with CS-1008 and paclitaxel/carboplatin versus placebo and paclitaxel/carboplatin | 1 year
Difference in objective response rate (ORR) of patients treated with CS-1008 and paclitaxel/carboplatin versus placebo and paclitaxel/carboplatin | 1 year
Difference in duration of response of patients treated with CS-1008 and paclitaxel/carboplatin versus placebo and paclitaxel/carboplatin | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Zentrum fur Pneumologie und Thoraxchirurgie, Grobhansdorf, Grobhansdorf
  - Asklepios Fachkliniken Munchen Gauting, Gauting

REFERENCES:
- [Derived] Reck M, Krzakowski M, Chmielowska E, Sebastian M, Hadler D, Fox T, Wang Q, Greenberg J, Beckman RA, von Pawel J. A randomized, double-blind, placebo-controlled phase 2 study of tigatuzumab (CS-1008) in combination with carboplatin/paclitaxel in patients with chemotherapy-naive metastatic/unresectable non-small cell lung cancer. Lung Cancer. 2013 Dec;82(3):441-8. doi: 10.1016/j.lungcan.2013.09.014. Epub 2013 Oct 1. PMID 24148258